CLINICAL TRIAL: NCT07110597
Title: Communicating Multiple Uncertainties Associated With the Benefits and Risks of New Cancer Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: Harvard Medical School / Harvard Pilgrim Health Care Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 540788 (study 2)
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Uncertainty; Prescription drug information
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Placebo Comparator): No information about uncertainty given.
  Interventions: Other: Control group
- 1 source of uncertainty (Experimental): Other: Statement communicating uncertainty with small magnitude of benefit
  Interventions: Other: Statement communicating 1 source of uncertainty
- 2 sources of uncertainties (Experimental): Other: Statements communicating uncertainty with a small magnitude of benefit and limited study population
  Interventions: Other: Statements communicating 2 sources of uncertainties
- 3 sources of uncertainties (Experimental): Other: Statements communicating uncertainty with a small magnitude of benefit, limited study population, and unvalidated surrogate endpoint
  Interventions: Other: Statements communicating 3 sources of uncertainties
- 4 sources of uncertainties (Experimental): Other: Statements communicating uncertainty with a small magnitude of benefit, limited study population, unvalidated surrogate endpoint, and limited study duration.
  Interventions: Other: Statements communicating 4 sources of uncertainties

INTERVENTIONS:
Other: Statement communicating 1 source of uncertainty — It is unknown whether patients with non-small cell lung cancer will notice an improvement with Zenova.
  Arms: 1 source of uncertainty
Other: Statements communicating 2 sources of uncertainties — It is unknown whether patients with non-small cell lung cancer will notice an improvement with Zenova.
  Zenova has not been studied in patients similar to Alex (patients with her race and ethnicity). It is unknown whether Zenova will work and what harms it will have for patients like her.
  Arms: 2 sources of uncertainties
Other: Statements communicating 3 sources of uncertainties — It is unknown whether patients with non-small cell lung cancer will notice an improvement with Zenova.
  Zenova has not been studied in patients similar to Alex (patients with her race and ethnicity). It is unknown whether Zenova will work and what harms it will have for patients like her.
  Zenova has only been shown to shrink the size of tumors. It is unknown whether Zenova improves how patients feel or how long they live.
  Arms: 3 sources of uncertainties
Other: Statements communicating 4 sources of uncertainties — It is unknown whether patients with non-small cell lung cancer will notice an improvement with Zenova.
  Zenova has not been studied in patients similar to Alex (patients with her race and ethnicity). It is unknown whether Zenova will work and what harms it will have for patients like her.
  Zenova has only been shown to shrink the size of tumors. It is unknown whether Zenova improves how patients feel or how long they live.
  Since patients given Zenova were followed for a short time, the longer-term benefits and harms of taking Zenova are unknown.
  Arms: 4 sources of uncertainties
Other: Control group — No information about uncertainty
  Arms: Control group

SUMMARY:
This nationally representative randomized survey of US adults will evaluate the effect of using brief statements to communicate multiple different sources of uncertainties about the benefits and harms of new cancer drugs on participants' decisions.

DETAILED DESCRIPTION:
Many newer cancer drugs are approved before uncertainties with their underlying clinical trial evidence have been adequately studied, in turn making it difficult to accurately determine the drug's benefits and harms. Prescription drug information rarely communicates these uncertainties. In a nationally representative sample of US adults, this study will evaluate the effect of using brief statements to communicate multiple different sources of uncertainties about the benefits and harms of new cancer drugs on participants' decisions.

In the pre-intervention phase, participants will be given information about a hypothetical new drug approved for the treatment of non-small cell lung cancer. Participants will be asked how likely they would be to take the drug, and how certain they are that the drug will work. Participants will then be randomized with equal allocation to 1 of 5 groups. The control group will receive information about a new cancer drug's benefits and harms; the intervention groups will also be given brief statements about sources of uncertainties with the drug's evidence (1, 2, 3, or 4 sources of uncertainties). The post-intervention questions will re-assess participants' decision making, perceptions of uncertainty, emotions, understanding, and trust.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Adults fluent in English
* Adults residing in the United States

Exclusion Criteria:

* Participants who do not meet each of the 3 inclusion criteria
* Participants who initiated the first survey about communicating individual sources of uncertainties (verified using unique participant identifiers assigned by the survey company)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3184 (Actual)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Change in decisions | Immediately prior to and after the intervention.
  "Imagine you were Alex and diagnosed with non-small cell lung cancer. How likely are you to take the new drug, Zenova?"
  4-point Likert scale for decision-making: very likely; somewhat likely; somewhat unlikely; very unlikely

SECONDARY OUTCOMES:
Change in understanding | Immediately prior to and after the intervention.
  Please answer rate your agreement with the following statements:
  Zenova works better than other treatments for non-small cell lung cancer Zenova's longer-term benefits and harms are well known Zenova has been studied in patients that are similar to Alex (race and ethnicity) Zenova improves how patients feel or how long they live Zenova has a very large benefit for patients with non-small cell lung cancer
  4-point Likert scale for understanding: strongly disagree; somewhat disagree; somewhat agree; strongly agree.
Change in perception of uncertainty | Immediately prior to and after the intervention.
  "How certain are you that Zenova will work for Alex?"
  4-point Likert scale for perception of uncertainty: very uncertain; somewhat uncertain; somewhat certain; very certain.
Change in emotions | Immediately prior to and after the intervention.
  If you were Alex, how worried would you feel about taking Zenova?
  4-point Likert scale for worry: extremely worried; slightly worried; not very worried; not worried at all.
Trust | Immediately prior to and after the intervention.
  To what extent do you think the information about Zenova is trustworthy? 4-point Likert scale: not at all trustworthy; somewhat untrustworthy; somewhat trustworthy; very trustworthy.
  To what extent do you think the FDA, who approved Zenova and produced this information, is trustworthy? 4-point Likert scale: not at all trustworthy; somewhat untrustworthy; somewhat trustworthy; very trustworthy.
  Did learning about these uncertainties with Zenova make you more or less trusting of the FDA? 4-point Likert scale: less trusting, somewhat less trusting, somewhat more trusting, more trusting.

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Economics and Political Science, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is the second of 2 studies on communicating uncertainties associated with the benefits and risks of new cancer drugs — https://www.clinicaltrials.gov/study/NCT06997185?term=communicating%20risk&viewType=Table&rank=8

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT07110597/Prot_SAP_ICF_000.pdf